CLINICAL TRIAL: NCT04211129
Title: Effect of Acupuncture on Crohn's Disease Via the Regulation of Trp-kyn Metabolism in Brain-gut Axis
Brief Title: Effect of Acupuncture on Patients With Crohn's Disease in Remission
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funds.
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Collaborators: Fudan University (Other); Ruijin Hospital (Other); Shanghai Mental Health Center (Other); Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZYS2019-02
Record Dates: First submitted 2019-12-22; First posted 2019-12-26 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Crohn Disease; Inflammatory Bowel Diseases
Keywords: acupuncture; Crohn's disease; brain functional activity
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture group (Experimental): Receiving acupuncture and moxibustion
  Interventions: Other: acupuncture
- sham acupuncture group (Sham Comparator): Receiving sham acupuncture and sham moxibustion
  Interventions: Other: Sham acupuncture

INTERVENTIONS:
Other: acupuncture — Patients receiving acupuncture and mild moxibustion, whom were treated 3 times per week for 12 weeks and followed up for 36 weeks. CV12 and Bilateral ST37, SP6, SP4, LR3, KI3, LI4 and LI11 were selected for acupuncture and bilateral ST25 and ST36 were selected for moxibustion. Hwato acupuncture device was used to blind the subjects, and had the deqi sensation. The surface temperature of acupoints was maintained at 43℃± 1℃ for moxibustion.
  Arms: acupuncture group
Other: Sham acupuncture — Patients receiving sham acupuncture and sham mild moxibustion, whom were treated 3 times per week for 12 weeks and followed up for 36 weeks. CV12 and Bilateral ST37, SP6, SP4, LR3, KI3, LI4 and LI11 were selected for acupuncture and bilateral ST25 and ST36 were selected for moxibustion. Same Hwato acupuncture device was used to blind the subjects, but do not puncturing into the skin and do not have the deqi sensation. The surface temperature of acupoints was maintained at 37℃± 1℃ for moxibustion.
  Arms: sham acupuncture group

SUMMARY:
To observe the therapeutic effect of acupuncture on Crohn's disease in remission and its influence of brain functional activity

DETAILED DESCRIPTION:
1. Effect of acupuncture on symptoms （functional gastrointestinal symptoms, Fatigue, insomnia, depression, anxiety and perceived stress）of CD
2. Effect of acupuncture on brain functional activity of CD

ELIGIBILITY:
Inclusion Criteria:

1. aged 16-70;
2. patients in remission (CDAI < 150);
3. patients were not taking medication or were only taking one or more of the following drugs: [prednisone ≤15mg/d, azathioprine (≤1mg/kg/d), methotrexate (≤15mg/w) or mesalazine (≤4g/d)] and prednisone was used for at least 1 month, while azathioprine, methotrexate or mesalazine was used for at least 3 months;
4. those who did not use TNF alpha and other preparations within 3 months before entering the study;
5. those who have never experienced acupuncture;
6. patients signing informed consent.

Exclusion Criteria:

1. patients who are recently pregnant or in pregnancy or lactation;
2. patients with serious organic diseases;
3. patients diagnosed as psychosis;
4. patients who take antibiotics, probiotics, traditional Chinese medicine and other drugs at the same time, or who suffer from multiple diseases and need to take other drugs for a long time, and may affect the observation of the efficacy of this trial;
5. severe skin diseases (such as erythema nodosum, pyoderma gangrenosum, etc.), eye diseases (such as iritis, uveitis, etc.), thromboembolic diseases and other serious extraintestinal manifestations;
6. there are serious intestinal fistula, abdominal abscess, intestinal stenosis and obstruction, perianal abscess, gastrointestinal hemorrhage, intestinal perforation and other complications;
7. patients with short bowel syndrome who have undergone abdominal or gastrointestinal surgery in the past half a year;
8. there are skin diseases or defects in the selected area of acupuncture and moxibustion that cannot be performed.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Brief Fatigue Inventory (BFI-C) | Week 12
  The mean change in BFI-C from baseline. The higher the score, the worse the condition. Greater than 0, the upper limit is 90.

SECONDARY OUTCOMES:
Brief Fatigue Inventory (BFI-C) | Week 24,52
  The mean change in BFI-C from baseline. The higher the score, the worse the condition. Greater than 0, the upper limit is 90.
The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) | Week 12, 24,52
  The mean change in FACIT-F from baseline. The higher the score, the worse the condition. The score range from 0 to 52.
Crohn's disease activity index （CDAI）score | Week 12, 24,36,48,52
  The mean change in CDAI from baseline. The higher the score, the worse the condition. Greater than 0, no upper limit.
Inflammatory bowel disease questionnaire (IBDQ) | Week 12, 24 and 52
  The mean change in IBDQ from baseline. The higher the score, the worse the condition.The score is range from 32 to 224.
Hospital anxiety and depression scale (HADS) | Week 12, 24 and 52
  The mean change in HADS from baseline. The higher the score, the more serious the disease. The depression and anxiety score is range from 0 to 21.
Patient Health Questionnaire Depression Scale (PHQ-9) | Week 12, 24 and 52
  The mean change in PHQ-9 from baseline. The higher the score, the more serious the disease. The depression and anxiety score is range from 0 to 27.
Generalized Anxiety Disorder (GAD-7) | Week 12, 24 and 52
  The mean change in gad-7 from baseline. The higher the score, the more serious the disease. The depression and anxiety score is range from 0 to 21.
The proportion of recurrences | Week 52
  Defined as CDAI > 150 and increase ≥ 70 points or need to adjust drug to control disease condition.
Brain functional and structural changes | Week 12
  measured by functional MRI
Colonoscopy or small bowel MR evaluation | Week 52
  measured by colonoscopy (SES-CD score) or small bowel MR (MaRIA score)
Laboratory tests | Week 12, 24, 36, and 52
  Serum C-reactive protein (CRP), erythrocyte sedimentation rate (ESR) and platelet count (PLT)

CONTACTS AND LOCATIONS:
Overall Officials: Huangan Wu, MD, PhD, Study Chair — Shanghai Research Institute of Acupuncture and Meridian
Locations (2):
- China (2):
  - Shanghai Research Institute of Acupuncture and Meridian, Shanghai
  - Yueyang Hospital of Integrated Traditional Chinese and Western medicine, Shanghai university of traditional Chinese medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No